CLINICAL TRIAL: NCT04348019
Title: Mealtime Matters: An 8-wk Randomized-Controlled Trial to Examine the Effects of a Daily Time-Restricted Feeding Protocol on Diet Quality
Brief Title: Effects of a Daily Time-Restricted Feeding Protocol on Diet Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associate Dean, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRF-DQ
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Diet, Healthy; Weight Change, Body; Dyslipidemias; Blood Pressure
Keywords: time restricted feeding; fasting; diet quality; body mass index; cardiometabolic biomarkers
MeSH Terms: conditions — Body Weight Changes; Dyslipidemias; Intermittent Fasting; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: 8-week randomized-controlled, 2-arm parallel design trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted feeding (Experimental): Participants in the intervention arm of the study will consume food and beverages of their choice within one hour of waking and the feeding window will extend 6 hours. Beyond these hours, participants will observe a prolonged fast (i.e., an 18-h overnight fast).
  Interventions: Behavioral: Fasting
- Control (Placebo Comparator): Participants in the control arm of the study will fast each night for 8 hours.
  Interventions: Behavioral: Fasting

INTERVENTIONS:
Behavioral: Fasting — Fasting was defined as no foods or caloric beverages.

SUMMARY:
As a result of unhealthful lifestyle practices including nighttime ingestion and excess energy-dense food and beverage intake, college students are presenting with metabolic abnormalities and excess weight gain that increases their risk for chronic health conditions including cardiovascular diseases and type 2 diabetes. Research has shown that prolonging nightly fasting intervals can result in health improvements in both animal models and human subjects. Time-restricted feeding (TRF), a form of intermittent fasting may offer an exciting, non-pharmacologic approach to improve cardiometabolic health in this population by restricting food intake to feeding windows that align with circadian biology.

DETAILED DESCRIPTION:
This 8-wk randomized-controlled, parallel arm trial will examine the effects of a daily 18 h fast (TRF protocol) compared to a daily 8-h (CON protocol) on (1) diet quality, (2) cardiometabolic health, and (3) anthropometry in college students enrolled at ASU. Institutional Review Board (IRB) approval will be granted prior to recruitment and commencement of trial activities. Participants will be stratified by age, waist circumference, gender, and METS (activity score) and randomly assigned to one of two study arms: intervention and control. [Women will begin the trial within 5 days of menses.] Participants in the intervention arm of the study will consume food and beverages of their choice within one hour of waking and the feeding window will extend 6 hours. Beyond these hours, participants will observe a prolonged fast (i.e., an 18-h overnight fast). Participants in the control arm of the study will fast each night for 8 hours. During fasting hours, participants will only be permitted to consume non-caloric beverages (preferably water only but unsweetened and non-caloric coffee, tea, etc. will be permitted). Participants will adhere to their daily protocol for 8 weeks. Participants will not receive diet instruction other than 'to fast' and are told to maintain their typical physical activity patterns for the duration of the trial. Participants will choose one 'cheat-day' per week where they are excused from the fasting protocols; this day of the week will be consistent throughout the 8-week trial. Diet quality will be measured by the REAP-S questionnaire, 24-h recalls will be obtained by a registered dietitian via a three-step multiple-pass interview method, a registered nurse or radiology technician will obtain fasting blood draws for biomarkers, and trained research personnel will obtain measures of anthropometry.

ELIGIBILITY:
Inclusion Criteria:

* healthy (no unresolved medical condition)
* non-smoking (includes vaping)
* normal to under-active (< 420 minutes of activity/week; not training for or competing in sports events)
* college students (≥18 years old)
* free of acute illnesses or diagnosed chronic diseases (by self-report)
* waist circumference ≥ 80 cm for women, and ≥ 94 cm for men. Participants will not be excluded based on race/ethnicity or socioeconomic status.

Exclusion Criteria:

* participants who regularly fast for >12 hours/d or adhere to a fasting regimen (i.e., alternate day fasting, Ramadan-style fasting, 5:2 fasting) at the time of screening or within the past six months
* those with weight loss attempt(s) or weight change (≥ 5 lbs.) within the past six months (including pregnancy)
* those with a history of weight cycling (repeated weight loss and weight gain over time)
* those who currently work night-shifts (i.e., midnight to 6AM), and those unwilling to adhere to the protocol will be excluded from the trial
* pregnant or lactating women, and women not on prescription contraceptives (i.e., birth control pills, IUDs, and patches) (however, if a female applicant states her menstrual cycle is regular, the need to be on prescription contraceptives will be waived)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Diet quality | Change from Baseline at week 8
  A REAP-S questionnaire will be completed for the previous week's intake during Trial Visits 1-3. The REAP-S questionnaire is a 16-item validated measure of diet quality whereby participants respond to questions that estimate the intake of fruits and vegetables, fiber, sugar, milk, fat, and dietary cholesterol. Responses of 'usually/often' will receive 1 point, 'sometimes' will receive 2 points, and 'rarely/never or does not apply to me' will receive 3 points. Per the REAP-S protocol, responses will be tabulated, and higher scores will indicate better diet quality.
Blood pressure | Change from Baseline at week 8
  Both systolic and diastolic blood pressure will be obtained prior to blood draw. Participants will be instructed to sit quietly with their feet planted flat on the floor. After a 10-minute rest period, a non-invasive Omron auto cuff blood pressure monitor equipped with IntelliSense technology, which allows the machine to inflate and deflate at optimum levels depending on arm size, will be utilized to obtain blood pressure in mm Hg.
Blood lipids | Change from Baseline at week 8
  . LDL and HDL cholesterol will be measured using a commercially available diagnostic test kit on a bench-top, fully automated, clinical chemistry analyzer (Randox Laboratories Ltd, Crumlin, UK), and results will be expressed in milligrams per deciliter (mg/dL). Triglycerides will be measured using a commercially available diagnostic test kit on a bench-top, fully automated, clinical chemistry analyzer (Randox Laboratories Ltd, Crumlin, UK), and results will be expressed in milligrams per deciliter (mg/dL).
Waist circumference | Change from Baseline at week 8
  Waist circumference will be obtained to the nearest 5 cm using a research-grade ergonomic measuring tape placed horizontally around participants' natural waist (i.e., narrowest circumference above the umbilicus). Waist circumference will be measured twice and averaged unless the difference between the first and second measurement is above 5 cm. In that event, a third measurement will be obtained, and the mean of the nearest two circumferences will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No